CLINICAL TRIAL: NCT02205437
Title: Novel Candidate Genes for Treatment Response to Antipsychotics in Schizophrenia: Evidence From Pharmacogenetics in the Light of Personalized Medicine
Brief Title: Novel Candidate Genes for Treatment Response to Antipsychotics in Schizophrenia
Acronym: GEXANT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Centro de Investigación Biomédica en Red de Salud Mental (Network); Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Benedicto Crespo-Facorro, Associate Professor of Psychiatry, Fundación Marques de Valdecilla
Other Study IDs: GEXANT
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2019-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Psychosis; Antipsychotics; Treatment response; Metabolic side effects; Gene expression; RNA; Genes
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Controls: Healthy subjects without psychotic disorder.
- Drug-naive patients: Drug-naive (never medicated) schizophrenia patients.
- Patients responder to treatment: Patients with a good clinical response to treatment (define by a marked improvement of positive symptoms) at 3 months and at 1 year.
- Patients non-responder to treatment: Patients with a poor clinical response to treatment at 3 months and at 1 year.
- Patients with metabolic side effects: Patients with metabolic side effects associated to treatment.
- Patients with non-metabolic side effects: Patients with no metabolic side effects associated to treatment.

SUMMARY:
Schizophrenia is a severe and chronic mental disorder. The lifetime risk of schizophrenia is around 1%. Its course is chronic and frequently disabling. The keystone of schizophrenia treatment is antipsychotic medications. The use of antipsychotics represents a huge public health and economic burden to society. Most of antipsychotics drugs are "metoo" drugs, directly or indirectly replicating dopamine D2 receptor blockade. Pharmaceutical companies have aimed to produce drugs with a general indication for all patients with schizophrenia with a "one-size-fits-all" strategy with no targeting or stratification. Second generation antipsychotics partly improve positive symptoms and are quite often associated to weight gain, metabolic changes and increased risk of cardiovascular diseases. Antipsychotics only achieve a certain degree of clinical improvement in a percentage of patients (45%) and 30% of the patients are treatment resistant. In light of the current deadlock, there is an urgent need to expand the horizon of pharmacological research by elucidating new mechanisms related to antipsychotic actions. An alternative strategy is the comparison of gene expression profiles in drug-naive accurately ill patients before and after antipsychotic treatment has been initiated. Our research group has a great experience in the field and has been working on this hypothesis in the latest years. We propose a continuation project to thoroughly explore the clinical implications (clinical response to antipsychotic drugs or emergence of metabolic side effects) of the variants in gene expression we have recently described in schizophrenia patients. This project takes advantage of an exceptional (regarding to the detailed knowledge of clinical outcome and side effect profile) longitudinal cohort of drug-naive patients with schizophrenia who had been followed up for three years at the University Hospital Marqués de Valdecilla.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed up for 3 years in the First Episode Psychosis Clinical Program (PAFIP).
* 15-60 years.
* Living in the catchment area.
* Experiencing their first episode of psychosis.
* No prior treatment with antipsychotic medication or, if previously treated, a total life time of adequate antipsychotic treatment of less than 6 weeks.
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for brief psychotic disorder, schizophreniform disorder, schizophrenia, or schizoaffective disorder.

Exclusion Criteria:

* Meeting DSM-IV criteria for drug dependence.
* Meeting DSM-IV criteria for mental retardation.
* Having a history of neurological disease or head injury.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals included in the First Episode Psychosis Clinical Program (PAFIP) at the University Hospital Marqués de Valdecilla (Santander - Cantabria).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement. | 1 year.
  Changes in the total scores of the Scale for the Assessment of Positive Symptoms (SAPS) and Negative Symptoms (SANS), the Brief Psychiatric Rating Scale (BPRS) and the severity scale of the Clinical Global Impression (CGI) scale.

SECONDARY OUTCOMES:
Changes in metabolic parameters. | 1 year.
  This parameters are Cholesterol, Triglycerides, Glucose and Homeostasis model assessment (HOMA) index.
Effect of gender and cannabis use in the profile of gene expression associated with schizophrenia. | 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo-Facorro, Professor, Principal Investigator — University Hospital Marqués de Valdecilla, IDIVAL, Department of Psychiatry, School of Medicine, University of Cantabria, Santander, Spain. CIBERSAM Centro Investigación Biomédica en Red Salud Mental, Madrid, Spain
Locations (1):
- University Hospital Marques de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No